CLINICAL TRIAL: NCT04800406
Title: Marginal Bone Height Changes Around Two Different Surface Treated Dental Implants Supporting Mandibular Complete Overdenture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Elboraey, Associate Professor, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16007
Record Dates: First submitted 2021-03-13; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Assess Marginal Bone Height Changes Around Dental Implants
Keywords: Implant surface treatment; Marginal bone height; Cone beam computed tomography
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Ten completely edentulous patients aged from 50-60 years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Dental Implants — Resorbable blast media surface treated dental implant and Acid etched surface treated dental implant.

SUMMARY:
Patients participating in this study were rehabilitated by mucosa supported maxillary complete denture and mandibular overdenture supported by two different surface treated implants; resorbable blast media (RBM) on the right and Acid etched on the left; retained by ball attachments. The marginal bone height changes around RBM and acid etched surface treated dental implants retaining mandibular complete overdenture were assessed by cone beam computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Free from any systemic diseases affecting the bone metabolism.
* Healthy, firm covering mucosa which is free from any signs of Inflammation or ulceration.
* Residual alveolar ridge with adequate height and width.
* Angel's class I classification maxillo - mandibular relationship.
* Sufficient inter arch space

Exclusion Criteria:

* Smoker.
* Patients with parafunction habits (clenching or bruxism).

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Marginal Bone height changes | one year
  The marginal bone changes around each type of dental implant were assessed by cone beam computed tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided